CLINICAL TRIAL: NCT00130572
Title: Randomized Placebo-Controlled Clinical Pilot Trial Regarding the Efficacy of Elidel Cream on Erosive Oral Lichen Planus
Brief Title: Efficacy of Elidel Cream on Erosive Oral Lichen Planus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CASM981CDE12
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Lichen Planus, Oral
MeSH Terms: conditions — Lichen Planus, Oral | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Pimecrolimus

SUMMARY:
The purpose of this study is to investigate whether topical applied pimecrolimus will lead to improvement of erosive oral lichen planus. This effect will be monitored by reduction of erosive mucosal area and reduction of patient's pain symptoms.

DETAILED DESCRIPTION:
Oral lichen planus is a mucosal inflammatory disease of unknown origin. It can be very painful especially if erosions appear on the oral mucosa.

In this study the efficacy of pimecrolimus compared to placebo in treatment of erosive oral lichen planus will be investigated. To this end the subjective pain and the amount of affected mucosa will be monitored before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and histologically confirmed diagnosis of erosive oral lichen planus
* Spontaneous or meal related oral pain
* No topical therapy 2 weeks prior to study start
* No systemic therapy 4 weeks prior to study start
* Signed informed consent

Exclusion Criteria:

* Pregnant or breast-feeding women
* Known allergy to macrolide antibiotics
* Known current active malignant disease or in patient's history
* Known immunodeficiency or HIV infection
* Participation at another clinical trial within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2004-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Reduction of a symptom score consisting of involved mucosal area and appearance of pain before and after treatment

SECONDARY OUTCOMES:
Patient's and investigator's global assessment after 4 and 8 weeks
Pimecrolimus blood level after 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tilo Biedermann, Prof. Dr. med., Principal Investigator — University of Tuebingen, Department of Dermatology
Locations (1):
- University Hospital, Department of Dermatology, Tübingen, Germany